CLINICAL TRIAL: NCT00731471
Title: A Phase I Study Evaluating the Safety and Immunogenicity of a New TB Vaccine, MVA85A, in Healthy Volunteers Who Are Infected With HIV
Brief Title: A Phase I Study of a New Tuberculosis (TB) Vaccine, MVA85A, in Healthy Volunteers With HIV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Centre Hospitalier Universitaire Le Dantec, Dakar, Senegal (Unknown)
Responsible Party: Dr Helen McShane, University of Oxford
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TB019
Record Dates: First submitted 2008-08-06; First posted 2008-08-11 (Estimated); Last update posted 2011-03-28 (Estimated); Status verified 2011-03

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — MVA 85A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 12 Healthy adults infected with HIV
  Interventions: Biological: MVA85A
- 2 (Experimental): 12 HIV+ adults on antiretroviral therapy
  Interventions: Biological: MVA85A

INTERVENTIONS:
Biological: MVA85A — Modified vaccinia virus Ankara expressing antigen 85A from Mycobacterium tuberculosis. Both arms will receive two vaccinations six months apart.

SUMMARY:
This is an open Phase I study of a candidate TB vaccine, MVA85A, in healthy subjects who are infected with HIV. It is designed to study the safety and immunogenicity of the vaccine.

DETAILED DESCRIPTION:
This study is designed to evaluate the safety of MVA85A in healthy volunteers in Senegal who are infected with HIV. In phase I studies, a single vaccination with MVA85A, when administered at a dose of 5 x 107pfu intradermally, has been shown to be safe in both mycobacterially naïve individuals, those previously vaccinated with BCG and latently infected individuals. We will use 1 x 10^8 pfu MVA85A intradermally in this study. A trial in BCG vaccinated subjects showed that the higher dose (1 x 10^8 pfu MVA85A) induced a significantly higher immune response but did not have a higher AE profile. In addition, because of a variable immune response, the trial in HIV positive subjects in the UK is split into two groups, the first getting 5 x 10^7 pfu and the second getting 1 x 10^8 pfu MVA85A. It has, therefore, been decided to use the higher dose in order to maximise the immune response whilst maintaining a good safety profile.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 50 years
* Resident in or near Dakar for the duration of the study
* Willingness to allow the investigators to discuss the volunteer's medical history with the volunteer's HIV lead physician
* Willing to use effective contraception throughout duration of study (if female)
* HIV antibody positive; diagnosed at least 6 months previously
* CD4 count >300
* Arm 1: HIV viral load not >100,000 copies per millilitre
* Arm 2: Undetectable HIV viral load
* Written informed consent

Exclusion Criteria:

* Any clinically significant abnormal finding on screening biochemistry or haematology blood tests or on urinalysis
* Group 1 only: Any ARV therapy within the past 6 months
* Previous history of TB disease and/or treatment
* Any AIDS defining illness
* Group 1: CD4 count nadir <300
* Group 2: CD4 count nadir <100
* CXR showing TB or evidence of other active infection
* Prior receipt of a recombinant MVA or Fowlpox vaccine
* Use of any investigational or non-registered drug, live vaccine or medical device other than the study vaccine within 30 days preceding dosing of study vaccine, or planned use during the study period
* Administration of chronic (defined as more than 14 days) immunosuppressive drugs or other immune modifying drugs within six months of vaccination. (For corticosteroids, this will mean prednisolone, or equivalent, ≥ 0.5 mg/kg/day. Inhaled and topical steroids are allowed.)
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, e.g. egg products
* Presence of any underlying disease that compromises the diagnosis and evaluation of response to the vaccine (including evidence of cardiovascular disease, history of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ), history of insulin requiring diabetes mellitus, any ongoing chronic illness requiring ongoing specialist supervision (e.g., gastrointestinal), and chronic or active neurological disease)
* History of > 2 hospitalisations for invasive bacterial infections (pneumonia, meningitis)
* Suspected or known current drug and/or alcohol abuse
* Seropositive for hepatitis B surface antigen (HBsAg) and/ or hepatitis C (antibodies to HCV)
* Evidence of serious psychiatric condition
* Any other on-going chronic illness requiring hospital specialist supervision
* Any confirmed or suspected immunosuppressive or immunodeficient condition, other than HIV infection, such as asplenia
* Evidence of hepatomegaly
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* Pregnant/lactating female and any female who is willing or intends to become pregnant during the study
* Any history of anaphylaxis in reaction to vaccination
* PI assessment of lack of willingness to participate and comply with all requirements of the protocol, or identification of any factor felt to significantly increase the participant's risk of suffering an adverse outcome

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2008-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Safety of MVA85A | Six months

SECONDARY OUTCOMES:
Immunogenicity of MVA85A | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Helen McShane, Principal Investigator — University of Oxford; Souleymane Mboup, Principal Investigator — Centre Hospitalier Universitaire Le Dantec
Locations (1):
- Centre Hospitalier Le Dantec, Dakar, Senegal

REFERENCES:
- [Derived] Dieye TN, Ndiaye BP, Dieng AB, Fall M, Brittain N, Vermaak S, Camara M, Diop-Ndiaye H, Ngom-Gueye NF, Diaw PA, Toure-Kane C, Sow PS, Mboup S, McShane H. Two doses of candidate TB vaccine MVA85A in antiretroviral therapy (ART) naive subjects gives comparable immunogenicity to one dose in ART+ subjects. PLoS One. 2013 Jun 28;8(6):e67177. doi: 10.1371/journal.pone.0067177. Print 2013. PMID 23840618